CLINICAL TRIAL: NCT02269995
Title: Post-marketing Surveillance of DC Bead in Patients With Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: DCB01S
Record Dates: First submitted 2014-08-22; First posted 2014-10-21 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular; Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- E7040
  Interventions: Device: E7040

INTERVENTIONS:
Device: E7040 — E7040 of optimal particle size (-300 um, 300-500 um, or 500-700 um to fit in a target vessel, target lesion, or embolized area) as transcatheter study device will be administered .
  Other Names: DC Beads

SUMMARY:
This surveillance's objectives are:

1. Unknown adverse reactions
2. Incidences of adverse drug reaction
3. Factors considered to have effect to safety and effectiveness

ELIGIBILITY:
Inclusion criteria:

Patients with Hepatocellular carcinoma

Exclusion criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-12-25 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by Adverse Events | Up to 30 days

SECONDARY OUTCOMES:
Efficacy of DC bead as assessed by embolic performance | Up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Background] Jpn J Intervent Radiol. 2017;32:136-141.